CLINICAL TRIAL: NCT03967340
Title: PREdiction of Chronic LUng Allograft Dysfunction
Acronym: PRELUD
Status: Active, not recruiting | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC18_0351
Record Dates: First submitted 2019-05-22; First posted 2019-05-30 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Lung Transplant Rejection
Keywords: chronic lung allograft dysfunction; lung transplantation; biomarkers; personalized medecine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood and serum will be collected and retained in a biorepository
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Lung transplant

SUMMARY:
Chronic lung allograft dysfunction (CLAD) is the leading cause of long-term mortality after lung transplantation. Several risk factors for CLAD have been identified, but the exact pathophysiology and triggering molecular factors remain largely unknown. Moreover, in clinical practice, no integration of the different risk factors is achieved. CLAD is therefore diagnosed most often late with the persistent decline in respiratory function, revealing a profound and irreversible alteration of the pulmonary graft. Several blood biomarkers that can predict the occurrence of CLAD more than 6 months before clinical diagnosis have been identified and validated. From these preliminary results, a composite score is being developed from independent samples from the COLT (COhort in Lung Transplantation) cohort. The main objective of this project is to validate this robust and predictive composite score (biological and clinical) of CLAD.

ELIGIBILITY:
Inclusion Criteria:

* Patients to receive lung transplants awaiting registration on the transplant waiting list
* Patients affiliated to a social security system
* Patients who have given their informed consent
* Patients weighing more than 26 kg
* Patients over 16 years of age

Exclusion Criteria:

* Pregnant or breastfeeding women
* Patients unable to follow the protocol
* Patients with concomitant inflammatory diseases, regardless of acute, chronic or infectious rejection.
* Patients with a history of cancer in remission for less than 5 years, with the exception of localized skin cancers, excluding melanoma.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients newly enrolled on the waiting list in transplant centres will be included in the PRELUD study.
  Based on the number of annual transplants in France (300/year), we plan to include 240 patients at the time of their registration on the transplant waiting list. Of these 240 patients, we estimate that 190 patients will be transplanted.
  It will be possible to include patients in emergencies. In this case, the consent of a trusted person or relative will be obtained and then the patient will give his or her consent as soon as his or her condition permits.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2020-09-10 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
MMP-9 levels in plasma, gene expression and lymphocyte levels in blood associated with Chronic Lung Allograft Dysfunction (CLAD) | 3 years

SECONDARY OUTCOMES:
Expression of the 3 genes BLK, POU2AF1 and TCL1A in whole blood associated with CLAD | 3 years
MMP-9 levels over time associated with CLAD | 3 years
Transitional B lymphocytes rate over time associated with CLAD | 3 years
T lymphocytes levels over time associated with CLAD | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Adrien TISSOT, Dr, Principal Investigator — Nantes University Hospital
Locations (10):
- France (10):
  - CHU de Bordeaux, Bordeaux
  - CHU de Grenoble, Grenoble
  - Centre Chirurgical Marie Lannelongue, Le Plessis-Robinson
  - CHU de Lyon, Lyon
  - AP-HM, Marseille
  - CHU de Nantes, Nantes
  - Hôpital Bichat, Paris
  - CHRU de Strasbourg, Strasbourg
  - Hôpital Foch, Suresnes
  - CHU de Toulouse, Toulouse